CLINICAL TRIAL: NCT01238783
Title: Safety and Efficacy of AL-15469A 0.5% / AL-6515 0.3% Ophthalmic Suspension for Treatment of Bacterial Conjunctivitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-061
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AL-15469A 0.5% and AL-65150.3% Ophthalmic Suspension (Experimental)
  Interventions: Drug: AL-15469A 0.5% and AL-6515 0.3% Ophthalmic Suspension
- AL-15469A 0.5% (Experimental)
  Interventions: Drug: AL-15469A 0.5%
- AL-6515 0.3% (Experimental)
  Interventions: Drug: AL-6515 0.3%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AL-15469A 0.5% and AL-6515 0.3% Ophthalmic Suspension — Topical ocular dosed 3 times per day for 3 days
  Arms: AL-15469A 0.5% and AL-65150.3% Ophthalmic Suspension
Drug: AL-15469A 0.5% — Topical ocular dosed 3 times per day for 3 days
  Arms: AL-15469A 0.5%
Drug: AL-6515 0.3% — Topical ocular dosed 3 times per day for 3 days
  Arms: AL-6515 0.3%
Drug: Vehicle — Topical ocular dosed 3 times per day for 3 days
  Arms: Vehicle

SUMMARY:
To assess safety and efficacy of AL-15469A 0.5% /AL-6515 0.3% Ophthalmic Suspension for treatment of bacterial conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any race
* 5 years of age and older at the time of the Day 1 visit
* with a primary clinical diagnosis of bacterial conjunctivitis.

Exclusion Criteria:

* Onset of bacterial conjunctivitis (signs and symptoms) more than 4 days
* Presence of punctal plug or punctal occlusion
* Visual Acuity worse than 20/80
* Upper respiratory infection

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Sustained Clinical Cure rate | Day 3
End of therapy Clinical Cure rate | Day 4

SECONDARY OUTCOMES:
Sustained bulbar conjunctival injection | Day 3
Microbiological Success | Day 4